CLINICAL TRIAL: NCT07003867
Title: Ventilator Inspiratory Trigger Sensitivity Adjustment Versus Threshold Device Training on Pulmonary Functions in Acute Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Zaytoonah University of Jordan (Other)
Responsible Party: Principal Investigator, Mohamed Saied Zidan, Assistant prof dr, Al-Zaytoonah University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB # 1/4/2024-2025
Record Dates: First submitted 2025-05-23; First posted 2025-06-04 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Ventilated Patients; Acute Stroke Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group ( threshold inspiratory muscle training ) (Active Comparator)
  Interventions: Other: Ventilator inspiratory trigger sensitivity adjustment , threshold device training
- Experimental group ( Adjustment of ventilator trigger sensitivity ) (Experimental)
  Interventions: Other: Ventilator inspiratory trigger sensitivity adjustment , threshold device training

INTERVENTIONS:
Other: Ventilator inspiratory trigger sensitivity adjustment , threshold device training — Ventilator inspiratory trigger sensitivity adjustment threshold device training

SUMMARY:
Neurological dysfunction is a common condition necessitating prolonged mechanical ventilation (PMV). Among patients with acute neurological diseases, 17% to 33% are intubated and mechanically ventilated for respiratory failure. Patients with acute neurological diseases requiring MV generally have adverse outcomes with a hospital mortality rate among patients with such diseases has been reported to be in the range of 16-33%. Inspiratory muscle weakness is common in patients receiving mechanical ventilation, especially patients with prolonged duration of mechanical ventilation. Inspiratory muscle training could limit or reverse these unhelpful squeal and facilitate more rapid and successful weaning.Hence, the importance of physical therapy emerged in helping patients to be weaned from ventilators by using various methods to strengthen the respiratory muscles in different ways.

DETAILED DESCRIPTION:
Mechanical ventilation (MV) is a life-saving intervention used worldwide in an estimated 15 million patients annually. Although70% of patients in intensive care units wean without difficulty on the first attempt, approximately 30% require prolonged weaning. Prolonged mechanical ventilation is associated with an increased risk of death ,poor long-term functional outcomes, and markedly higher healthcare costsMechanical Ventilation (MV) is used to restore or enhance pulmonary gas exchange in patients who are unable to maintain adequate alveolar ventilation. Conditions that necessitate the use of MV include but are not restricted to neuromuscular diseases, respiratory failure secondary to chronic obstructive lung disease and following surgery with general anesthesia . A high proportion of patients who require prolonged MV for more than 48 hours do not survive for 1 year, and those who survive have a significantly reduced functional status and quality of life . Prolonged MV has a detrimental impact on the diaphragm, and this has been termed as Ventilator-Induced Diaphragmatic Dysfunction (VIDD ).Inspiratory muscle training is a type of training in which the patient inhales against resistive loads or pressure threshold-loads while the expiration is unloaded, that applies a load to the diaphragm and accessory inspiratory muscles to increase their strength and endurance .The trigger phase corresponds to the process in which the patient's spontaneous breathing triggers the ventilator to work. The inhalation phase corresponds to the process in which PAW rises to the plateau pressure while maintaining pressure support

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40-60 years.
* Diagnosed with acute stroke patients.
* Body mass index (BMI) 18:35 kg/m².
* conscious oriented patients with Glasgow coma score ≥ 13.
* PH>7.25 and arterial oxygen saturation >90%

Exclusion Criteria:

* Persistent hemodynamic instability as life threatening arrhythmias, acute heart failure, angina.
* Severe breathlessness when spontaneously breathing.
* Any progressive neuromuscular disease that would interfere with responding to inspiratory muscle training.
* Spinal cord injuries.
* Skeletal pathology (scoliosis, flail chest, spinal instrumentation) that would seriously impair the movement of the chest wall and ribs.
* Patients on heavy sedation and respiratory muscle paralysis

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-06-10 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Pulmonary compliance ( mL/cmH2O ) | pre and post 1 week
  A measure of the lung expandability, which is important in ideal respiratory system function. It refers to the ability of the lungs to stretch and expand. Lung compliance can be calculated by dividing volume by pressure (C = V/P), Pulmonary compliance was assessed daily in all mechanically ventilated patients using data obtained directly from the ventilator system (CARESCAPE -R860/USA)

SECONDARY OUTCOMES:
Paco2 (mmHg) | pre and post 1 week of intervention
  partial pressure of carbon dioxide in arterial blood , using Blood Gas analyzer:(Abbott Laboratories Pharmaceutical Company, Singapore)
PaO2 ( mmHg ) | pre and post 1 week of intervention
  partial pressure of oxygen in arterial blood ,using Blood Gas analyzer:(Abbott Laboratories Pharmaceutical Company, Singapore)
HCO3 ( mEq/L ) | Pre and post 1 week of intervention
  Refers to bicarbonate, a key component of the blood's acid-base balance ,using Blood Gas analyzer:(Abbott Laboratories Pharmaceutical Company, Singapore)
pH | Pre and post 1 week of intervention
  Refers to the acidity or alkalinity of the blood ,using Blood Gas analyzer:(Abbott Laboratories Pharmaceutical Company, Singapore)

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Saied Zidan, Cairo, Egypt